CLINICAL TRIAL: NCT05463731
Title: Assessment of Safety, Tolerability, and Efficacy Measured by Amyloid Reduction of LY3372993 in Early Symptomatic Alzheimer's Disease
Brief Title: A Study of Remternetug (LY3372993) in Participants With Alzheimer's Disease (TRAILRUNNER-ALZ 1)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18467; J1G-MC-LAKC (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-07-14; First posted 2022-07-19 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
Keywords: Mild cognitive impairment; Alzheimer's disease; Dementia; Amyloid-beta therapy; Amyloid Plaque; Disease modifying
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The main treatment period is double-blinded and the addendum is open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Remternetug (IV) (Experimental): Participants will receive remternetug intravenously (IV)
  Participants will receive remternetug IV during the treatment period, then switch to placebo IV in the extension period.
  Interventions: Drug: Remternetug (IV)
- Remternetug (SC) (Experimental): Participants will receive one of two dosing regimens of remternetug subcutaneously (SC)
  Participants will receive remternetug SC during the treatment period, then switch to placebo SC in the extension period.
  Interventions: Drug: Remternetug (SC)
- Placebo (Placebo Comparator): Participants will receive placebo matching remternetug IV or SC.
  Participants will receive placebo IV during the treatment period, then switch to remternetug IV in the extension period.
  Participants will receive placebo SC during the treatment period, then switch to LY3372993 SC in the extension period.
  Interventions: Drug: Placebo
- Open-Label Addenda Remternetug (IV) (Experimental): Participants will receive one of six dosing regimens of remternetug IV during the open-label addenda.
  Interventions: Drug: Remternetug (IV)
- Open-Label Addenda Remternetug (SC) (Experimental): Participants will receive one of nine dosing regimens of remternetug SC during the open-label addenda.
  Interventions: Drug: Remternetug (SC)

INTERVENTIONS:
Drug: Remternetug (IV) — Administered IV
  Other Names: LY3372993
  Arms: Open-Label Addenda Remternetug (IV); Remternetug (IV)
Drug: Remternetug (SC) — Administered SC
  Other Names: LY3372993
  Arms: Open-Label Addenda Remternetug (SC); Remternetug (SC)
Drug: Placebo — Administered IV or SC
  Arms: Placebo

SUMMARY:
The reason for this study is to collect safety and efficacy information regarding the study drug remternetug in participants with early symptomatic Alzheimer's disease (AD).

DETAILED DESCRIPTION:
TRAILRUNNER-ALZ 1 is a Phase 3, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of remternetug in participants with early symptomatic AD. Initially, 600 participants will enroll in the double-blind treatment period. Participants in the double-blind treatment period will receive remternetug or placebo administered via subcutaneous injection or intravenous infusion.

Following the 52-week main study period, participants will continue participation for up to an additional 76 weeks in an extension period. Participants who previously received remternetug will receive placebo and participants who previously received placebo will receive remternetug. Thus, all participants will receive remternetug if they complete the study.

An additional 974 participants with early Alzheimer's disease will be enrolled to an addendum safety cohort. The participants will be administered open label remternetug via subcutaneous injection or intravenous infusion. Participants enrolled into the addendum safety cohort are not eligible for the extension period.

ELIGIBILITY:
Inclusion Criteria:

* Gradual and progressive change in cognitive function ≥6 months prior to screening.
* A Mini-Mental (MMSE) score of 20 to 30 (inclusive) at screening.
* Has an amyloid PET scan result consistent with the eligibility criteria.
* Have a reliable study partner who will provide written informed consent to participate and is in frequent contact with the participant.
* Have adequate literacy, vision, and hearing for the neuropsychological testing in the opinion of the investigator at the time of screening.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Males and females will be eligible for this study.
* Women not of childbearing potential (WNOCBP) may participate in this trial.

Exclusion Criteria:

* Current serious or unstable illnesses that, in the investigator's opinion, could interfere with the analyses in this study; or has a life expectancy of <24 months.
* History of cancer with high risk of recurrence and preventing completion of the trial.
* Participants with any current primary psychiatric diagnosis other than AD that in the investigator's opinion, is likely to confound interpretation of the drug effect, affect cognitive assessment, or affect the participant's ability to complete the study.
* History of clinically significant multiple or severe drug allergies.
* Have any clinically important abnormality at screening, as determined by investigator that could be detrimental to the participant, could compromise the study, or show evidence of other etiologies for dementia.
* Screening magnetic resonance imaging (MRI) which shows evidence of significant abnormality that would suggest another potential etiology for progressive dementia or a clinically significant finding that may impact the participant's ability to safely participate in the study.
* Have any contraindications for MRI or positron emission tomography (PET).
* Have had prior treatment with a passive anti-amyloid immunotherapy.
* Have received active immunization against Aβ in any other study.
* Have known allergies to remternetug related compounds, or any components of the formulation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1667 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Reach Amyloid Plaque Clearance on Amyloid PET Scan for Remternetug versus Placebo | Week 52

SECONDARY OUTCOMES:
Mean Absolute Change from Baseline in Brain Amyloid Plaque on Amyloid PET Scan for Remternetug versus Placebo | Baseline, Week 52
Percentage of Participants Who Reach Amyloid Plaque Clearance on Amyloid PET Scan for Remternetug versus Placebo | Week 24
Mean Absolute Change from Baseline in Brain Amyloid Plaque on Amyloid PET Scan for Remternetug versus Placebo | Baseline, Week 24
Time to Reach Complete Amyloid Plaque Clearance on Remternetug versus Placebo | Up to Week 52
Pharmacokinetics (PK) Observed Trough Serum Concentration (Cmin) of Remternetug | Baseline to Week 52
Number of Participants with Treatment Emergent Anti-Drug Antibodies (TE-ADAs) | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (76):
- United States (73):
  - MD First Research - Chandler, Chandler, Arizona
  - Hope Clinical Research, Inc., Canoga Park, California
  - North County Neurology Associates, Carlsbad, California
  - Wr- Pri, Llc, Encino, California
  - Neuro-Pain Medical Center, Fresno, California
  - Irvine Clinical Research, Irvine, California
  - Kaizen Brain Center, La Jolla, California
  - Anderson Clinical Research, Redlands, California
  - Mountain Neurological Research Center, Basalt, Colorado
  - Alpine Clinical Research Center, Boulder, Colorado
  - Colorado Springs Neurological Associates, Colorado Springs, Colorado
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Ki Health Partners, LLc, dba New England Institute for Clinical Research, Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - VIN-Julie Schwartzbard, Aventura, Florida
  - Brain Matters Research, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Encore Research Group- Jacksonville Center for Clinical Research, Jacksonville, Florida
  - ClinCloud - Maitland, Maitland, Florida
  - K2 Medical Research, Maitland, Florida
  - ClinCloud - Viera, Melbourne, Florida
  - Merritt Island Medical Research, LLC, Merritt Island, Florida
  - VIN-Andrew Lerman, Miami, Florida
  - Optimus U Corporation, Miami, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research - Winter Park, Orlando, Florida
  - Emerald Coast Neurology - Airport Boulevard, Pensacola, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Alzheimer's Research and Treatment Center, Stuart, Florida
  - Brain Matters Research, Stuart, Florida
  - Tallahassee Neurological Clinic, Tallahassee, Florida
  - Charter Research - Lady Lake, The Villages, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Columbus Memory Center, PC, Columbus, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Great Lakes Clinical Trials - Andersonville, Chicago, Illinois
  - AMITA Health - Alexian Brothers Neurosciences Institute Clinical Research, Elk Grove Village, Illinois
  - Covenant Medical Center, Waterloo, Iowa
  - Cotton O'Neil Clinical Research Center - Central Office, Topeka, Kansas
  - Care Access - Lake Charles, Lake Charles, Louisiana
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Citizens Memorial Hospital District, Bolivar, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of New Jersey, Toms River, New Jersey
  - Neurological Associates Albany, Albany, New York
  - AMC Research, Matthews, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - Valley Medical Research, Centerville, Ohio
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Center for Cognitive Health, Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Keystone Clinical Studies, Plymouth Meeting, Pennsylvania
  - Rhode Island Mood & Memory Research Institute, East Providence, Rhode Island
  - Neurology Clinic, P.C., Cordova, Tennessee
  - Texas Diabetes & Endocrinology, P.A., Austin, Texas
  - Gadolin Research, Beaumont, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Re:Cognition Health, Fairfax, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Universal Research Group, Tacoma, Washington
- Japan (3):
  - Memory Clinic Toride, Toride, Ibaraki
  - Katayama Medical Clinic, Kurashiki, Okayama-ken
  - Memory Clinic Ochanomizu, Bunkyo-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Remternetug (LY3372993) in Participants With Alzheimer's Disease (TRAILRUNNER-ALZ 1) — https://trials.lilly.com/en-US/trial/351135